CLINICAL TRIAL: NCT01418651
Title: Efficacy and Safety of Milnacipran in the Treatment of Fibromyalgia in an Elderly Population: an Open-label Study
Brief Title: Efficacy and Safety of Milnacipran in the Treatment of Fibromyalgia in an Elderly Population
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of subjects
Sponsor: Banner Health (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sandra Jacobson MD - Research Physician, Banner Sun Health Research Inst.
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-007
Record Dates: First submitted 2011-03-28; First posted 2011-08-17 (Estimated); Last update posted 2011-08-17 (Estimated); Status verified 2011-01

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Milnacipran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Milnacipran (Experimental): Drug
  Interventions: Drug: Savella

INTERVENTIONS:
Drug: Savella — milnacipran 25 to 200 mg daily, divided into two doses (morning and evening)

SUMMARY:
Participants will undertake a 12-week, open-label study of milnacipran in a well-characterized cohort of patients with fibromyalgia syndrome (FMS) who are 65 years and older to investigate the short-term efficacy and safety of this drug in the elderly population. The investigators hypothesize that milnacipran will be effective in treating fibromyalgia syndrome (FMS), and will be prove to be safe when patients are selected for the absence of pre-existing blood pressure abnormalities and other serious medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients.
* Age 65 years or older.
* Fibromyalgia diagnosed according to ACR 1990 criteria.
* Pain Score ≥ 10 on Gracely scale at screening and baseline assessments.
* Discontinuation of other dual-acting antidepressant medications, including duloxetine, venlafaxine, and tricyclic antidepressants for a period not less than 4.5 times the drug half-life as of the baseline evaluation.

Exclusion Criteria:

* Uncontrolled hypertension (BP ≥ 140/90) at screening or baseline evaluations.
* Baseline orthostasis (documented drop in SBP ≥ 20 mmHg or in DBP ≥ 10 mmHg within 3 minutes after standing) at screening or baseline evaluations.
* Psychosis, active suicidality, current episode of major depression or other severe psychiatric illness, or current alcohol/substance abuse or dependence as assessed by the MINI.
* Significant cardiovascular disease, including atrial fibrillation or other dysrhythmia, congestive heart failure, valvular heart disease, or QTc prolongation on baseline EKG (> 450 msec).
* Uncontrolled narrow angle glaucoma.
* History of seizures.
* Use of MAO inhibitor drugs within the last 14 days.
* Abnormal baseline liver or renal function tests.
* Dementia or other syndrome of cognitive impairment that could interfere with the subject's ability to participate fully in the assessment protocol.
* Obstructive uropathy in males.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Change in self-reported severity of pain over 12 weeks of treatment in persons aged 65 and older | 14 months
  Percent change in self-reported severity of pain (averaged Visual Analog Scale scores) over 12 weeks of treatment.
  Rate of occurrence of adverse events necessitating drug discontinuation

SECONDARY OUTCOMES:
Determine the effects of milnacipran on cognition | 14 months
  Change in functional activity (FIQ), perceived health (SF-36), and severity of pain (Gracely scale).
  Incidence and severity of treatment-emergent adverse events. Change in sleep quality and daytime sleepiness as measured by the Pittsburgh Sleep Quality Index and Epworth Sleepiness Scale.
  Change in other sleep/wake parameters(actigraphy measures). Change in cognitive test scores from baseline to the 12 week visit. Patient global impression of change score.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Jacobson, MD, Principal Investigator — Banner Health
Locations (1):
- Banner Sun Health Research Institute, Sun City, Arizona, United States